# CONSENT FORM AND AUTHORIZATION FOR DISCLOSURE OF PROTECTED HEALTH INFORMATION

# STUDY TITLE: A DOUBLE-BLIND, RANDOMIZED STUDY TO COMPARE ONABOTULINUMTOXIN A VS. TRIAMCINOLONE FOR INTRAVAGINAL TRIGGER POINT INJECTIONS IN THE TREATMENT OF CHRONIC PELVIC PAIN

Principal Investigator: Jamie Bartley, DO

Address: 3601 West 13 Mile Road, Royal Oak, MI 48073

Hospital: William Beaumont Hospital, Royal Oak

#### INTRODUCTION

#### Why is this study being done?

You are being asked to participate in a clinical research study. The purpose of clinical research is to look at the nature of disease and try to develop improved methods to diagnose and treat disease. The doctor or clinician in charge of the study believes you meet the initial requirements to take part in the study. Before agreeing to participate, it is important for you to read and understand the following explanation of the research procedures. This Consent and Authorization form describes the purpose, procedures, benefits, risks and discomforts of the study. It also describes the alternatives available to you, and your right to withdraw (quit) from the study at any time.

Dr. Kenneth Peters, one of the doctors conducting this study at William Beaumont Hospital, has received payments from Allergan, the company that makes the study drug, for consulting.

Please read this information carefully and ask as many questions as you like before deciding whether or not you would like to take part in this research study.

The goal of this study is to compare the effectiveness of two different medications used in intralevator (pelvic) trigger point injections (injections into extremely painful areas of a muscle) to treat chronic pelvic pain. We are comparing onabotulinumtoxinA (BOTOX®) (a drug prepared from the bacterial toxin botulin which temporarily paralyzes muscles) to triamcinolone (Kenalog) (a synthetic corticosteroid used as an anti-inflammatory agent).

A total of 40 patients will take part in the study here at William Beaumont Hospital, Royal Oak.

# How long will I be in the study?

If you decide to take part in this study, your participation is expected to last approximately six months. You may not take part in this study if you are currently enrolled in another related research study which could alter or influence the study results.

IRB NUMBER: 2015-008 IRB APPROVAL DATE: 12/05/2017 IRB EXPIRATION DATE: 11/29/2018

#### **DESCRIPTION OF THE STUDY**

# What will happen if I take part in the research study?

You are being asked to take part in this research study because you have been diagnosed with chronic pelvic pain with trigger points. Chronic pelvic pain has been described as long lasting, non-cyclical pain that occurs below the umbilicus. Trigger points are knot-like bands of muscle that cause pain when touched.

If you agree to take part in this study you will be randomly assigned to one of two treatment groups. Randomization is like "the flip of a coin." Double-blinded means that neither you nor your study doctor will know which medication you receive. In case of an emergency, the treatment can be unblinded to determine which therapy you have received. You will be randomized to receive either onabotulinumtoxinA with ropivacaine (a "numbing" medication) or triamcinolone with ropivacaine for your trigger point injection.

The following will occur at the specified study visits:

# **Screening Evaluation and Treatment**

The study will be explained to you in detail, and you will have as much time as you need to ask questions. You will be asked to read and sign this Consent and Authorization form before any study-related procedures are performed. The following tests and procedures should be done to determine if you qualify to participate in this study:

- Review of your medical history, including an assessment of your last menstrual period and contraceptive use. Review of medications you are currently taking and medications that you have taken in the past
- A pregnancy test if you are of child-bearing potential
- A vaginal examination will be performed by the study clinician to confirm the presence of high tone pelvic floor dysfunction (too much tension) and to determine that you do not have vaginitis (an inflammation or infection in the vagina). Vaginal pH and wet mount (sample of vaginal discharge) will be performed. If you have vaginitis you will be given a prescription for the appropriate medication. You may be re-screened 3 days after treatment. Also, a "Q-tip test" is performed. A Q-tip (cotton swab) is used to lightly test the vaginal area for pain and tenderness. Completion of guestionnaires about your pain
- Vital signs (blood pressure, pulse, respirations)

You will be eligible for full enrollment into the study after consenting to study participation, completing all screening evaluations, and meeting all entry criteria. The intralevator trigger point injections may occur at this visit or you may return to the clinic within 7 to 14 days to have the treatment.

There will be six injections in the vaginal/pelvic floor area: 1, 3, 5, 7, 9, and 11 o'clock. A tampon will then be inserted for approximately 5 minutes. You will be monitored for any side effects for a minimum of 30 minutes after the treatment. You will be given an ice pack to place on the treatment area, warm blankets and water or juice if you would like. Your vital

signs will be taken and you will be asked to give a pain score prior to your discharge from the clinic.

#### One month follow-up visit

You will return to the clinic approximately 30 days after the treatment and the following activities will take place:

- Review of your medical history, including an assessment of your last menstrual period and contraceptive use. Review of medications you are currently taking and medications that you have taken in the past
- Evaluation of any new medical events that have occurred since your last visit
- A vaginal examination to determine that you do not have vaginitis (an inflammation or infection in the vagina). Vaginal pH and wet mount (sample of vaginal discharge) will be performed. If you have vaginitis you will be given a prescription for the appropriate medication. Also, a "Q-tip test" is performed. A Q-tip (cotton swab) is used to lightly test the vaginal area for pain and tenderness. The study doctor will also assess your pain at the trigger point(s).
- Completion of questionnaires about your pain
- Vital signs (blood pressure, pulse, respirations)

The study doctor will review your treatment results with you and discuss if any additional treatment will begin. Permitted treatments include physical therapy, vaginal valium, and repeat trigger point injections. Triamcinolone will be used for the injections, but you will not be given onabotulinumtoxinA to prevent overdose of onabotulinumtoxinA. If onabotulinumtoxinA injections are advised, you would be withdrawn from the study and un-blinded.

#### Three month follow-up visit

You will return to the clinic approximately 90 days after the treatment and the following activities will take place:

- Review of your medical history, including an assessment of your last menstrual period and contraceptive use. Review of medications you are currently taking and medications that you have taken in the past
- Evaluation of any new medical events that have occurred since your last visit
- A vaginal examination to determine that you do not have vaginitis (an inflammation or infection in the vagina). Vaginal pH and wet mount (sample of vaginal discharge) will be performed. If you have vaginitis you will be given a prescription for the appropriate medication. Also, a "Q-tip test" is performed. A Q-tip (cotton swab) is used to lightly test the vaginal area for pain and tenderness. The study doctor will also assess your pain at the trigger point(s).
- Completion of questionnaires about your pain
- Vital signs (blood pressure, pulse, respirations)

The study doctor will review your treatment results with you and discuss if any additional treatment will begin. Permitted treatments include physical therapy, vaginal valium, and repeat

IRB NUMBER: 2015-008 IRB APPROVAL DATE: 12/05/2017 IRB EXPIRATION DATE: 11/29/2018 intralevator trigger point injections. Triamcinolone will be used for the injections, but you will not be given onabotulinumtoxinA to prevent overdose of onabotulinumtoxinA. If onabotulinumtoxinA injections are advised, you would be withdrawn from the study and unblinded.

#### Six month follow-up visit

You will return to the clinic approximately 180 days after the treatment and the following activities will take place:

- Review of your medical history, including an assessment of your last menstrual period and contraceptive use. Review of medications you are currently taking and medications that you have taken in the past
- Evaluation of any new medical events that have occurred since your last visit
- A vaginal examination to determine that you do not have vaginitis (an inflammation or infection in the vagina). Vaginal pH and wet mount (sample of vaginal discharge) will be performed. If you have vaginitis you will be given a prescription for the appropriate medication. Also, a "Q-tip test" is performed. A Q-tip (cotton swab) is used to lightly test the vaginal area for pain and tenderness. The study doctor will also assess your pain at the trigger point(s).
- Completion of questionnaires about your pain
- Vital signs (blood pressure, pulse, respirations)

The study doctor will review your treatment results with you and discuss if any additional treatment will begin. Permitted treatments include physical therapy, vaginal valium, and repeat trigger point injections. Triamcinolone will be used for the injections, but you will not be given onabotulinumtoxinA to prevent overdose of onabotulinumtoxinA. If onabotulinumtoxinA injections are advised, you would be withdrawn from the study and un-blinded.

\* While in-person study visits are preferable, the follow up visits may be completed as a phone call visit, if the participant is otherwise unable or unavailable. The questionnaires will be collected via mail.

In the event the study visit cannot be completed in-person,

- You will receive a telephone call from the study staff to review medications you are currently taking and review any problems you may be experiencing.
- You will be sent the follow up questionnaires to complete and a self-addressed stamped envelope for questionnaire return

#### **FDA Clinical Trial Information**

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### PARTICIPANT RESPONSIBILITIES

You should maintain your normal daily activities or physical therapy programs during your participation in the research study. You should not start any new medications, therapies or exercise programs during the study. Tell a member of the study staff promptly if you start taking a new drug or change the dose of an existing drug (including any over-the-counter medications or herbal supplements).

You will be asked to note any side effects or medical problems you may experience while you are taking part in this study. For any illnesses or injuries, you should contact the study doctor immediately at the number listed on this Consent and Authorization form or in an emergency situation call 911 (or go to the nearest hospital emergency room).

# **RISKS, SIDE EFFECTS AND DISCOMFORTS**

Ask your physician what the standard of care risks are as well as the study risks. What side effects or risks can I expect from being in the study?

#### **Risks of Trigger Point Injections:**

#### Most Frequent (occurring more than 10% of the time):

- Slight discomfort during the vaginal exam
- Light bleeding at the trigger point injection site
- Pain during the trigger point injection

#### Rare (occurring less than 1% of the time):

- Vaginal hematoma (collection of blood in the tissue)
- Infection

#### Risks of onabotulinumtoxinA:

# **Less Frequent (occurring from 1% to 10% of the time):**

- Transient urinary retention (temporary inability to urinate)
- Transient flatal incontinence (temporary accidental passing of gas)
- Transient fecal incontinence (temporary accidental loss of stool)
- Slight temporary fatique

# Rare (occurring less than 1% of the time):

- Trouble talking
- Lower extremity weakness
- Lower extremity numbness

#### **Risks of triamcinolone:**

#### Rare (occurring less than 1% of the time):

- Headache
- Dizziness
- Weight gain

- Hyperglycemia (high blood sugar)
- Trouble sleeping

#### **Risks of ropivacaine:**

# Rare (occurring less than 1% of the time):

- Hypertension (high blood pressure)
- Hypotension (low blood pressure)
- Arrhythmia (abnormal heart rate)
- Tachycardia (rapid heart rate)
- Headache
- Rash
- Lower extremity weakness
- Urinary retention (inability to urinate)
- Urinary incontinence (accidental loss of urine)
- Local anesthetic toxicity (numbing medication could be absorbed through the bloodstream into the rest of the body affecting your breathing, heartbeat, blood pressure)

There is a risk of an allergic reaction from any medication. Symptoms may include swelling, skin rash and/or headache. Just to be safe, you should go to the nearest emergency room if you were to experience worsening or unexpected difficulty swallowing or talking, trouble breathing or muscle weakness. It is important to know that these symptoms can occur days to weeks after an injection of onabotulinumtoxinA. There may be unknown side effects or problems that could result in serious illness or even death.

There is a rare risk of breach of confidentiality (release of information which personally identifies you).

Not all possible effects are known. With any medication or therapy, unusual, unexpected or previously unreported side effects may occur. You will be informed of any significant new findings, which develop during the course of this research study which may change your decision to continue participating in this study.

# **Pregnancy Warning**

If you are a woman who is pregnant or becomes pregnant during the research study, there could be harmful effects to you or your unborn child. It is important you not be pregnant or breast-feeding during any time in this study. Women of childbearing potential must agree to use birth control. If you are a woman of childbearing potential you must have a negative pregnancy test before entering the study.

#### **BENEFITS**

# What are the benefits of taking part in this study?

There may be no direct benefit to you from taking part in this study. Your chronic pelvic pain may improve, but this cannot be guaranteed. Information gained from the results of this study may be of benefit to others in the future, with a similar medical condition.

IRB NUMBER: 2015-008
IRB APPROVAL DATE: 12/05/2017
IRB EXPIRATION DATE: 11/29/2018

#### **ALTERNATIVE OPTIONS**

#### What are my choices other than taking part in this study?

You do not have to take part in this study to receive treatment for your condition. If you do not choose to participate in the study, you can still get trigger point injections and participate in other treatments. Other treatments to decrease pain include the use of vaginal valium and pelvic floor physical therapy. The risks include:

# **Risks of Vaginal Valium:**

# Rare (occurring less than 1% of the time):

- Slight Temporary Fatique
- Hypotension
- Weakness
- Rash

# **Risks of Pelvic Floor Physical Therapy** Rare (occurring less than 1% of the time):

Temporary muscular pain

#### **ECONOMIC CONSIDERATIONS**

#### What are the costs of taking part in this study?

The study medications including onabotulinumtoxinA and triamcinolone (and ropivicaine) will be provided to you at no cost for your initial treatment visit. There will be no cost to you for the study procedures described in this Consent and Authorization form (for example, pregnancy test (1), and questionnaires (5)). Routine procedures you would have had done even if you were not taking part in this study will be billed to your health insurance company and/or group health plans as usual (for example, Q-tip test (4-5), vaginal exam (4-5), trigger point injection procedure (1-4), triamcinolone and ropivicaine used for additional trigger point injections at follow up visits (0-3)). If these routine care costs are not covered by your health insurance/group health plan, the cost will be your responsibility.

You will be reimbursed for your time and travel (etc.) during the course of the study. You will be paid a total of \$75 if you complete all of the study visits. A check for \$15.00 will be sent to you by William Beaumont Hospital approximately two weeks after the completion of each of the five study visits.

#### COMPENSATION

#### What happens if I am injured because I took part in this study?

Your involvement in this study is voluntary. The possible risks and side effects which might occur during the course of the research study have been described in this Consent and Authorization form.

A research injury is any physical injury or illness caused by the medications, devices, or procedures required by the study which are administered, used, or performed appropriately.

HIC #2015-008 Version # 8.23.2017

These medications, devices, or procedures are different from the medical treatment you would have received if you had not taken part in the study.

Should you experience a research injury, there are no designated funds provided for subsequent medical care or compensation by either the study doctor/clinician or William Beaumont Hospital.

#### What are my rights if I take part in this study?

You are not giving up any of your legal rights by signing this form.

# CONFIDENTIALITY, DISCLOSURE AND USE OF YOUR INFORMATION Will my medical information be kept private?

In order for this research study to take place, you must also authorize the researchers to access and use some of your protected health information (PHI). PHI is information which could identify you as an individual such as name, address, date of birth, etc. By signing this Consent and Authorization Form, you give William Beaumont Hospital permission to use and/or disclose (release) your health information related to this research. Your medical and billing records collected for the purpose of the study will remain confidential, but may be disclosed (released) or used by the following and/or their representatives:

- The investigators (study doctor/clinician, research staff)
- William Beaumont Hospital
- The Food and Drug Administration
- Other governmental regulatory agencies (domestic and/or foreign)
- Your health insurance company and/or group health plans and their intermediaries (companies contracted to process claims) may also have access to your medical and billing records of the study.
- Primary Care Physician

## **Optional Notification to the Primary Physician**

The research doctor would like to inform your primary physician of your participation in the research study. If you agree, we will need you to give us the name of the primary physician to allow us to contact them.

| Yes, I want the stud | y doctor to inform my Primary Care Physician/Specialist of my |
|---|---|
| · | he study doctor to inform my Primary Care Physician/Specialist of my |
| I do not have a Prir | mary Care Physician/Specialist<br>my Primary Physician/Specialist |
| <br>Participant's Initials | <br>Date |

**IRB EXPIRATION DATE: 11/29/2018** 

The purpose for this disclosure (release) or use is, for example, to assure compliance with the study protocol, to evaluate the effectiveness of the study, and/or to provide protection to you as a research study participant. The disclosure and use of your information will continue after your involvement in the study has ended. There is no expiration date for the use of your medical and billing records from the study. Any information about you disclosed to the parties identified above may be re-disclosed by them; however, such re-disclosure is not under the protections of this Consent and Authorization.

You will not be identified in any publication or other release of study results, data, and other information (such as in professional writings, at professional meetings, and in the study sponsor's product information, and/or advertising or other promotional materials).

If you decide to withdraw your authorization for the researchers to access and use your personal health information before the end of the study, you will be withdrawn from the research study. However, where the study relied on your Consent and Authorization for the time you participated in the study, your Consent and Authorization cannot be withdrawn and the information already collected may still be used and disclosed as you previously authorized.

# STOPPING STUDY PARTICIPATION

# What if I decide to stop taking part in the study?

Taking part in this research study is completely voluntary. You may choose not to take part or to stop being in the study (withdraw) at any time without penalty or loss of benefits to which you are otherwise entitled, or without jeopardizing your medical care by your physician at William Beaumont Hospital. However, if you do not agree to sign this Consent and Authorization form, you will not be able to take part in this study.

If you decide to withdraw from the study you will need to notify the study doctor/clinician, in writing, of your decision to stop taking part in the study. This notice may be sent to Dr. Jamie Bartley at William Beaumont Hospital, 3601 West 13 Mile Road, Royal Oak, MI 48073.

Your participation in this study may be stopped by the study doctor/clinician or study sponsor, without your consent, for any reason, which will be explained to you. Examples include:

- The study medication or procedures appear to be medically harmful to you.
- You fail to follow directions for participating in the study.
- It is discovered you do not meet the study requirements.
- The study is canceled.
- It is determined to be in your best interest (for example, your disease has progressed despite treatment).

If your study doctor/clinician stops your participation, or you decide not to continue, you may be asked to have a final study visit or examination, in order for you to be discontinued from the study in a safe and orderly manner.

#### **CONTACTS**

#### Who can answer my questions about the study?

You may talk to the study doctor/clinicians about any questions or concerns regarding your study participation, or you think you may have suffered a research-related injury. The doctor/clinician in charge of the study, Dr. Jamie Bartley, may be reached at: 248-898-0898 to answer your questions.

Your contact person is Amanda Schonhoff, RN. You may contact her at 248-551-1225.

If you have questions regarding your rights as a research participant, or have problems, concerns, complaints, want information or would like to offer input, you may contact the Institutional Review Board (Human Investigation Committee) Chairperson at (248) 551-0662. The Human Investigation Committee is charged with the oversight of all human participant research conducted at William Beaumont Hospital facilities.

**IRB NUMBER: 2015-008** 

HIC #2015-008 Version # 8.23.2017

## STATEMENT OF VOLUNTARY PARTICIPATION

I have read the above, have asked questions and have received answers about this study to my satisfaction. I understand what I have read and willingly give my consent to participate in **A DOUBLE-BLIND, RANDOMIZED STUDY TO COMPARE ONABOTULINUMTOXIN A VS. TRIAMCINOLONE FOR INTRAVAGINAL TRIGGER POINT INJECTIONS IN THE TREATMENT OF CHRONIC PELVIC PAIN.** I understand I will receive a signed copy of this document and will be promptly informed of any new findings regarding this study. I further authorize the use or disclosure of my health and personal information contained in records as described above.

| RESEARCH PARTICIPANT NAME (PLEASE PRINT) | | |
|---|---|---|
| RESEARCH PARTICIPANT SIGNATURE | DATE | TIME |
| ALTERNATIVE SIGNATURE (IF RESEARCH PARTIC<br>AS THE PERSONAL/LEGAL REPRESENTATIVE OF THE ST<br>PARTICIPANT SECTION, AND CHECK ONE OF THE BOXE<br>AUTHORIZATION: | TUDY PARTICIPANT, PLEASE PRINT | |
| <del></del> | ABLE POWER OF ATTORNEY EY LETTER MUST BE PRESENT & VERIFIED B | NEXT OF KIN Y 2 PHYSICIANS |
| NAME (PLEASE PRINT) | RELATIONSHIP | TO PARTICIPANT |
| SIGNATURE | DATE | TIME |
| WITNESS TO SIGNATURE ON COI | NSENT WITNESS TO CO | NSENT PROCESS AND SIGNATURE |
| WITNESS NAME (PLEASE PRINT) | | |
| WITNESS SIGNATURE | DATE | TIME |
| <b>AUTHORIZED CONSENT PROVIDE</b> I have explained this study and have offe discussion or clarification. | _ | n opportunity for any furthe |
| NAME (PLEASE PRINT) | CREDENTIALS | PHONE NUMBER |
| <br>SIGNATURE | DATE | TIME |

IRB NUMBER: 2015-008